CLINICAL TRIAL: NCT05077306
Title: Effect of Musical Listening on Anxiety and Depression in Patients Hospitalized for Covid-19: a Randomized Controlled Trial
Brief Title: Receptive Music Therapy on Anxiety and Vital Parameters in Hospitalized Covid-19 Patients.
Acronym: MADC-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Prof.Nicola Brienza, professor, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID.MT
Record Dates: First submitted 2021-10-08; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV2 Infection
Keywords: music therapy; anxiety; stress; quality of life; vital parameters
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy group (Experimental): Patients receive an individual single session of receptive music therapy in presence.
  Interventions: Other: music therapy group
- Control group (No Intervention): Patients receive standard care

INTERVENTIONS:
Other: music therapy group — individual bedside single session of receptive music therapy (RMT) by a certified Music therapist- GIM fellow in presence. STAI Y-1 was administered 5 min. before session (STAI Y-1 PRE) and 15 min. after session (STAI Y-1 POST) in paper form. HR and O2Sat were recorded from the bedside monitor 3 times: start session (T0), 10 min. (T1), end session (T2).Participants i were asked to fill in an optional open-ended question concerning their experience with music therapy.
  Arms: music therapy group

SUMMARY:
Hospitalized patients for Covid-19 are extremely isolated from their families for a long and uncertain period of time .This traumatic separation makes patients vulnerable to different degrees of stress disorders as well as depression and anxiety , fear of the unknown and dying, sleeplessness, agitation, discomfort, pain, immobility, frustration and inability to relax .

MusicTtherapy has been shown to play a valuable role in the care of patients with serious illness, helping to address physical symptoms and psychological distress .

The aim of this study was to evaluate the feasibility of introducing Music therapy (MT) on site with Covid-19 patients as a supporting complementary/non-pharmacological intervention, to investigate the immediate effects a single MT session has on anxiety, heart rate (HR), oxygen saturation (O2Sat) and satisfaction compared to standard care.

In order to verify the hypotheses of the study, an RCT (mixed-methods approach pre -post design) will be carried out on patients diagnosed with SARS-COV2 admitted to Covid Hospital Bari, randomized into two groups: control group (B) and treatment group (A). .

The study starts on 15th April 2021 and it is expected to run for 1 mounth (15th May 2021).

The study is funding by University of Bari.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* not severe neurological or psychiatric conditions
* not hearing impairment
* not intubated

Exclusion Criteria:

* age under 18 years
* severe neurological or psychiatric conditions
* hearing impairment
* intubated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory Y-1 | through study completion - an average of 30 days
  State Trait Anxiety Inventory Y-1(STAI-Y1) was used to measure how the subject felt in that moment. Subjects were asked to rate the intensity of their anxious feelings on 20 items on a four point scale: not at all, somewhat, moderately so, or very much so. STAI-Y values <40 defined absence of anxiety, between 40 and 50 mild anxiety, 51-60 moderate anxiety, and> 59 severe anxiety
State Trait Anxiety Inventory Y-1 | through study completion- an average of 30 days
  State Trait Anxiety Inventory Y-1(STAI-Y1) was used to measure how the subject felt in that moment. Subjects were asked to rate the intensity of their anxious feelings on 20 items on a four point scale: not at all, somewhat, moderately so, or very much so. STAI-Y values <40 defined absence of anxiety, between 40 and 50 mild anxiety, 51-60 moderate anxiety, and> 59 severe anxiety. T1-during session.
State Trait Anxiety Inventory Y-1 | through study completion - an average of 30 days
  State Trait Anxiety Inventory Y-1(STAI-Y1) was used to measure how the subject felt in that moment. Subjects were asked to rate the intensity of their anxious feelings on 20 items on a four point scale: not at all, somewhat, moderately so, or very much so. STAI-Y values <40 defined absence of anxiety, between 40 and 50 mild anxiety, 51-60 moderate anxiety, and> 59 severe anxiety. T2- end session

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Brienza, Phd, Principal Investigator — University of Bari
Locations (1):
- AOUC Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fallek R, Corey K, Qamar A, Vernisie SN, Hoberman A, Selwyn PA, Fausto JA, Marcus P, Kvetan V, Lounsbury DW. Soothing the heart with music: A feasibility study of a bedside music therapy intervention for critically ill patients in an urban hospital setting. Palliat Support Care. 2020 Feb;18(1):47-54. doi: 10.1017/S1478951519000294. PMID 31104642
- [Background] Mofredj A, Alaya S, Tassaioust K, Bahloul H, Mrabet A. Music therapy, a review of the potential therapeutic benefits for the critically ill. J Crit Care. 2016 Oct;35:195-9. doi: 10.1016/j.jcrc.2016.05.021. Epub 2016 May 28. PMID 27481759
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Result] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Derived] Giordano F, Losurdo A, Quaranta VN, Campobasso N, Daleno A, Carpagnano E, Gesualdo L, Moschetta A, Brienza N. Effect of single session receptive music therapy on anxiety and vital parameters in hospitalized Covid-19 patients: a randomized controlled trial. Sci Rep. 2022 Feb 24;12(1):3154. doi: 10.1038/s41598-022-07085-8. PMID 35210504